CLINICAL TRIAL: NCT05628922
Title: Response-adapted Modulation Therapy for Locally Advanced Nasopharyngeal Carcinoma Based on Circulating Epstein-Barr Virus DNA Level Post Induction Chemotherapy
Brief Title: Modulation Therapy for Locally Advanced NPC Based on Plasma EBV DNA Level Post-ICT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, M.D., Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Remodel 1.0
Record Dates: First submitted 2022-06-11; First posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Nasopharyngeal Cancer
Keywords: Epstein-Barr virus DNA; Immunotherapy; Programmed Cell Death 1 antibody; Induction chemotherapy
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — toripalimab; Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early Responders (Experimental): those with undetectable plasma EBV DNA after first cycle of induction chemotherapy (GP regimen)
  Interventions: Other: Induction chemotherapy and concurrent chemoradiation
- Intermediate Responders (Experimental): those with detectable plasma EBV DNA after first cycle of induction chemotherapy (GP regimen), and undetectable plasma EBV DNA at completion of induction chemotherapy
  Interventions: Drug: Toripalimab; Other: Induction chemotherapy and concurrent chemoradiation
- Late Responders (Experimental): those with detectable plasma EBV DNA after first cycle and at completion of induction chemotherapy (GP regimen)
  Interventions: Drug: Toripalimab; Other: Induction chemotherapy and concurrent chemoradiation

INTERVENTIONS:
Drug: Toripalimab — Early Responders: They receive the second and third cycle of induction chemotherapy (GP regimen), followed by cisplatin-based concurrent chemoradiation.
  Intermediate Responders: they received the second and third cycle of induction chemotherapy (GP regimen) with combination of toripalimap (240mg d1, q3w * 2 cycles), followed by cisplatin-based concurrent chemoradiation.
  Late responders: they received the second and third cycle of induction chemotherapy (GP regimen) with combination of toripalimap (240mg d1, q3w * 2 cycles), followed by cisplatin-based concurrent chemoradiation. At 4-6 weeks post-chemoradiation, they received adjuvant capecitabine and toripalimab for 6 months.
  Other Names: JS001
  Arms: Intermediate Responders; Late Responders
Other: Induction chemotherapy and concurrent chemoradiation — Induction chemotherapy (GP regimen) and cisplatin-based concurrent chemoradiation.
  GP regimen: Gemcitabine 1.0 g d1,d8, cisplatin 25mg/m2 d1-3 q3w Cisplatin based chemotherapy: cisplatin 80mg/m2 given in three consecutive days, q3w * 2 cycles.

SUMMARY:
Nasopharyngeal carcinoma is biologically different from traditional head and neck squamous cell carcinoma. The mainstay treatment for locally advanced nasopharyngeal carcinoma is cisplatin-based concurrent chemoradiation. Recent phase III randomized control trials have demonstrated that induction chemotherapy plus concurrent chemoradiation further improved progression-free survival.

However, not every patient has good response to induction chemotherapy. Evidence has accumulated that those with poor response to induction chemotherapy, or those with detectable Epstein-Barr Virus (EBV) DNA post induction chemotherapy, correlated with poorer progression-free survival. Huang CL et al. (Int J Radiat Oncol Bio Phys. 2019) reported that plasma EBV DNA load at completion of induction chemotherapy was an independent and earlier predictor for progression-free survival and overall survival in locally advanced nasopharyngeal carcinoma. Lv J et al. (Nat Commun. 2019) demonstrated that real-time monitoring of plasma EBV DNA response added prognostic information, and had the potential uitility for risk-adapted treatment intensification in nasopharyngeal carcinoma.

Therefore, investigators selects those with poor plasma EBV DNA response during and after induction chemotherapy, and intensifies the treatment with combination of anti-PD-1 antibody, in order to improve progression-free survival in locally advanced nasopharyngeal carcinoma, according to response-adapted strategy.

DETAILED DESCRIPTION:
In this study, investigators enroll patients with locally advanced nasopharyngeal carcinoma. All the patients recieve GP-based induction chemotherapy. After one cycle of induction chemotherapy, plasma EBV DNA and head and neck MR are performed.

Based on clinical efficacy and changes of plasma EBV DNA, patients with good response will directly receive concurrent chemoradiation (CCRT). Patients with intermediate response will be randomized to immunotherapy group (GP combined with toripalimab for two additional cycles then CCRT) and standard group (GP for two additional cycles then CCRT). Patients with poor response will be switched to TP regimen combined with toripalimab, followed by CCRT. The main endpoint is 2 year progression-free survival rate.

The aim of this study is to clarify whether response-adapted strategy based on clinical efficacy and EBV DNA response confers survival benefit to patients with locally advanced nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must sign the informed consent form, and must be willing and able to comply with the visits, treatment regimen, laboratory tests and other requirements specified in the study protocol;
2. Age at diagnosis: 18-70 years old;
3. Firstly diagnosed, pathologically confirmed primary nasopharyngeal carcinoma with "non-keratinizing carcinoma (WHO criteria)";
4. Locally advanced nasopharyngeal carcinoma (T3-4N0-1M0, TanyN2-3M0), staged according to the American Joint Committee on Cancer (AJCC) 8th edition clinical staging system;
5. Pretreatment EBV DNA >0;
6. ECOG score: 0-1 points;
7. Does not receive any treatment after the diagnosis of nasopharyngeal carcinoma;
8. Normal bone marrow function: white blood cell >4*109/L, neutrophil count >1.5*109/L, hemoglobin concentration > 90g/L, platelet count >100*109/L;
9. Normal liver and kidney function: total bilirubin ≤1.5 times the upper limit of normal; aspartate aminotransferase and/or alanine aminotransferase ≤ 2.5 times the upper limit of normal; creatinine clearance ≥ 60mL/min;
10. For those with hepatitis B infection, the HBV DNA load must be < 2500 copies/ml at the time of screening; For those with anti-hepatitis C virus antibody, HCV RNA must be negative at the time of screening;
11. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to use reliable contraception (e.g. condoms, regular contraceptives as directed) from screening through 1 year after treatment.

Exclusion Criteria:

1. Pathologically confirmed primary nasopharyngeal carcinoma with "keratinizing carcinoma or basaloid squamous cell carcinoma";
2. Previous or current other malignancy other than adequately treated non-melanoma skin cancer, carcinoma in situ of the cervix, and papillary thyroid carcinoma;
3. Pretreatment plasma EBV DNA undetectable;
4. History of radiation therapy prior to standard therapy (except for non-melanoma skin cancer, and the previous radiation field did not overlap with the current treatment for nasopharyngeal carcinoma);
5. Patients who received surgical treatment (except for diagnostic biopsy), biological therapy, chemotherapy or immunotherapy before enrollment;
6. Conditions mentioned below: 1) Currently enrolled in other interventional clinical trial; 2) Systemic hormonal or other immunosuppressive therapy with an equivalent dose of > 10mg prednisone/day within 28 days prior to informed consent; 3) Receipt of live vaccines within 30 days prior to enrollment; 4) Surgery or trauma within 30 days prior to enrollment;
7. Uncontrolled heart disease, such as :1) heart failure, NYHA ≥ 2; 2) unstable angina; 3) history of myocardial infarction within 1 year; 4) supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. History of stroke within 6 months;
9. Patients with severe active infection within 30 days prior to enrollment, that must be treated with systemic antibacterial, antifungal or antiviral therapy;
10. Active autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary disease, nephritis, vasculitis, hyperthyroidism, etc.). Except for type I diabetes, hypothyroidism requiring hormone replacement therapy, and vitiligo not requiring systemic treatment, inactive childhood asthma that does not require treatment as an adult;
11. Positive anti-HIV antibody or diagnosis of other innate or acquired immunodeficient, immunosuppressive disease, history of organ transplantation;
12. Interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy within 1 year;
13. Active tuberculosis infection, or previous lung tuberculosis infection within 1 year, or previous lung tuberculosis infection more than 1 year prior to enrollment but did not receive standard anti-tuberculosis treatment;
14. Positive hepatitis B surface antigen and hepatitis B virus DNA ≥ 2500 copies/ml or Positive hepatitis C RNA;
15. Pregnant or lactating women (pregnancy test should be considered for sexually active women of childbearing age);
16. Other conditions that may jeopardize patient safety or compliance as assessed by investigator, such as serious illness (including psychiatric disorders) requiring prompt treatment, severely abnormal test results, and other family or social risk factors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-07-02 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 year
  the time from the date of enrollment to progression of disease

SECONDARY OUTCOMES:
Overall survival | 2 year
  the time from the date of enrollment to death
Locoregional recurrence-free survival | 2 year
  the time from date of enrollment to locoregional recurrence
Distant metastasis-free survival | 2 year
  the time from date of enrollment to distant metastasis
Adverse effects | up to 2 year
  evaluated according to CTCAE 5.0 version
Quality of Life | up to 2 year
  evaluated according to EORTC QLQ-C30
Quality of Life | up to 2 year
  evaluated according to EORTC QLQ-H&N35

CONTACTS AND LOCATIONS:
Overall Officials: Chao-su Hu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No